CLINICAL TRIAL: NCT05276492
Title: Abiraterone Dose De-Escalation Study: A Prospective Study Evaluating Decreasing Dosing Regimens of Abiraterone 500 mg in Men With Prostate Cancer to Find Lowest Recommended Dose.
Brief Title: Decreasing Dosing Regimens of Abiraterone 500 mg in Men With Prostate Cancer to Find Lowest Recommended Dose.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed by PI due to not meeting primary endpoint
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB21-1869
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostate Neoplasm; Prostate Cancer Metastatic
Keywords: prostate cancer; prostate adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: Dose Regimen 1 (Experimental): You will be enrolled in the study based on the study group that is open at that particular time. If you are enrolled in this group, you will receive:
  - Abiraterone 500 mg and prednisone 5mg with a low-fat meal every other day.
  You will take 2 pills (500 mg total) of abiraterone acetate, first thing in the morning with breakfast. The tablets should be swallowed whole and not crushed, chewed, or dissolved in water. This breakfast should be a low-fat meal (avoid high calorie foods with a high percentage of fat, such as bacon or sausage). You will be asked to document the details of the meal/taking abiraterone in a daily log.
  You will also take prednisone 5 mg daily in the form of tablets taken by mouth with approximately 8 ounces of water with food. You do not have to take prednisone and abiraterone at the same time of day. If you inadvertently miss a dose of the study drug, you should take the dose the next day and record this on your Drug Diary.
  Interventions: Drug: Abiraterone Oral Tablet; Drug: Prednisone tablet; Other: Drug Dairy/Log; Drug: Low-fat meal
- Group 2: Dose Regimen 2 (Experimental): You will be enrolled in the study based on the study group that is open at that particular time. If you are enrolled in this group, you will receive:
  - Abiraterone 500 mg and prednisone 5mg with a low-fat meal on day 1, day 3, day 5 of every week
  You will take 2 pills (500 mg total) of abiraterone acetate, first thing in the morning with breakfast. The tablets should be swallowed whole and not crushed, chewed, or dissolved in water. This breakfast should be a low-fat meal (avoid high calorie foods with a high percentage of fat, such as bacon or sausage). You will be asked to document the details of the meal/taking abiraterone in a daily log.
  You will also take prednisone 5 mg daily in the form of tablets taken by mouth with approximately 8 ounces of water with food. You do not have to take prednisone and abiraterone at the same time of day. If you inadvertently miss a dose of the study drug, you should take the dose the next day and record this on your Drug Diary.
  Interventions: Drug: Abiraterone Oral Tablet; Drug: Prednisone tablet; Other: Drug Dairy/Log; Drug: Low-fat meal
- Group 3: Dose Regimen 3 (Experimental): You will be enrolled in the study based on the study group that is open at that particular time. If you are enrolled in this group, you will receive:
  - Abiraterone 500 mg and prednisone 5mg with a low-fat meal on day 1 and day 4 of every week
  You will take 2 pills (500 mg total) of abiraterone acetate, first thing in the morning with breakfast. The tablets should be swallowed whole and not crushed, chewed, or dissolved in water. This breakfast should be a low-fat meal (avoid high calorie foods with a high percentage of fat, such as bacon or sausage). You will be asked to document the details of the meal/taking abiraterone in a daily log.
  You will also take prednisone 5 mg daily in the form of tablets taken by mouth with approximately 8 ounces of water with food. You do not have to take prednisone and abiraterone at the same time of day. If you inadvertently miss a dose of the study drug, you should take the dose the next day and record this on your Drug Diary.
  Interventions: Drug: Abiraterone Oral Tablet; Drug: Prednisone tablet; Other: Drug Dairy/Log; Drug: Low-fat meal
- Group 4: Dose Regimen 4 (Experimental): You will be enrolled in the study based on the study group that is open at that particular time. If you are enrolled in this group, you will receive:
  - Abiraterone 500 mg and prednisone 5mg with a low-fat meal on day 1 of every week
  You will take 2 pills (500 mg total) of abiraterone acetate, first thing in the morning with breakfast. The tablets should be swallowed whole and not crushed, chewed, or dissolved in water. This breakfast should be a low-fat meal (avoid high calorie foods with a high percentage of fat, such as bacon or sausage). You will be asked to document the details of the meal/taking abiraterone in a daily log.
  You will also take prednisone 5 mg daily in the form of tablets taken by mouth with approximately 8 ounces of water with food. You do not have to take prednisone and abiraterone at the same time of day. If you inadvertently miss a dose of the study drug, you should take the dose the next day and record this on your Drug Diary.
  Interventions: Drug: Abiraterone Oral Tablet; Drug: Prednisone tablet; Other: Drug Dairy/Log; Drug: Low-fat meal

INTERVENTIONS:
Drug: Abiraterone Oral Tablet — Abiraterone is used in combination with prednisone to treat a certain type of prostate cancer that has spread to other parts of the body. Abiraterone is in a class of medications called androgen biosynthesis inhibitors. It works by decreasing the amount of certain hormones in the body.
  Other Names: Yonsa; Zytiga
Drug: Prednisone tablet — Prednisone is a corticosteroid (cortisone-like medicine or steroid). It works on the immune system to help relieve swelling, redness, itching, and allergic reactions.
  Other Names: Deltasone; Prednicot; Rayos; Sterapred; Sterapred DS
Other: Drug Dairy/Log — A drug dairy/log that will the study team will give for you to document information about the study drugs and meals you take during the study.
Drug: Low-fat meal — A low-fat meal that will be taken with abiraterone. If you have questions about what is considered "a low-fat" meal during the study, ask the study doctor or research staff.

SUMMARY:
Doctors leading this study plan to collect new information about the lowest effective dose of abiraterone acetate in study participants with prostate cancer who are taking abiraterone in combination with prednisone for the first time. The duration of this study will be about 3 months (12 weeks). How long you stay on abiraterone, and at what dose after completion of the 12 weeks of study drug administration, will be up to you and your treating physician.

DETAILED DESCRIPTION:
Doctors leading this study plan to collect new information about the lowest effective dose of abiraterone acetate in study participants with prostate cancer who are taking abiraterone in combination with prednisone for the first time. The duration of this study will be about 3 months (12 weeks). How long you stay on abiraterone, and at what dose after completion of the 12 weeks of study drug administration, will be up to you and your treating physician.

Therefore, this study will evaluate if alternative dosing strategies with 500 mg pills may be equally effective as taking abiraterone 1000 mg daily. This study will specifically assess whether taking 500 mg of abiraterone every other day with a low-fat meal, or 500 mg with a low-fat meal at less frequent intervals (fewer times per week), is equally effective in treating prostate cancer as the 1000 mg/day dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed prostate cancer with plans to initiate abiraterone acetate
* Have never received prior abiraterone or other androgen receptor modulators, including enzalutamide, apalutamide, or darolutamide.
* Must have a baseline DHEA-S level of >20 mg/dL (in order to adequately assess DHEA-S response)
* A minimum washout of 28 days for any other anticancer therapy other than medical or surgical castration, prior to first dose of study drug is required.
* Any other radiotherapy or radionuclide require 28-day washout prior to first dose of study drug.
* Denosumab or zoledronic acid are allowed.
* Eastern Cooperative Oncology Group performance status ≤ 2 (Appendix A).
* Participants must have normal hepatic function as defined by clinical lab values set by the study doctor/research team.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Therapy with other hormonal therapy, including any dose of megestrol acetate (Megace), finasteride (Proscar), dutasteride (Avodart), or any herbal product known to decrease Prostate-Specific Antigen levels or any systemic corticosteroid (other than prednisone ≤10mg/day) within 4 weeks prior to first dose of study drug.
* Inability to swallow capsules or known gastrointestinal malabsorption.
* Blood pressure that is not controlled despite > 2 oral agents (SBP >160 and DBP >90 documented during the screening period with no subsequent blood pressure readings <160/100).
* Serum K+ < 3.5 mmoL/L. Patients with a K+ < 3.5 mmoL/L are required to have a documented subsequent K+ >3.5 prior to enrollment to be eligible.
* Serious intercurrent infections or non-malignant medical illnesses that are uncontrolled.
* Active psychiatric illness/social situations that would limit compliance with protocol requirements.
* Serious heart issues/congestive heart failure as assessed by New York Heart Association's definition of class II, class III, or IV congestive heart failure.
* Taking other medications or drugs with strong inhibitors or inducers of CYP3A4 (See Section 8.12 below for list of strong inhibitor or inducers) due to concerning possible drug-drug interactions with abiraterone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-11-16 (Actual)

PRIMARY OUTCOMES:
Change in DHEA-S Levels Among Participants at 4 Weeks | 4 weeks
  Efficacy of different dosing regimens of abiraterone 500 mg as assessed by decrease/reduction in serum dihydroepiadrosterone sulfate (DHEA-S) levels among participants at 4 weeks.

SECONDARY OUTCOMES:
Change in Prostate-Specific Antigen (PSA) Levels of Participants at 12 Weeks | 12 weeks
  The effects of different dosing regimens of abiraterone 500 mg on serum as assessed by a reduction/decline in Prostate-Specific Antigen (PSA) levels (a 50% decline in PSA from baseline) at 12 weeks.
Rate of Adverse Events Reported Among Participants in Different Abiraterone Dosing Regimen Groups | 12 weeks
  Rate of adverse events reported among participants taking abiraterone 500 mg in different dosing groups as assessed by the Common Terminology Criteria for Adverse Events version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Szmulewitz, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States